CLINICAL TRIAL: NCT00803686
Title: A Randomized, Open-Label, Placebo-Controlled, Two-Period Crossover Study of the Effect on CTx-1 Concentrations of a Single 200 μg Recombinant Salmon Calcitonin (rsCT) Dose Given at Night to Normal, Healthy, Postmenopausal Women
Brief Title: A Study of Oral Calcitonin Given at Night to Healthy Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UGL-OR0803; Bio-Kinetic No.: 13808 (Other: Unigene Laboratories 0803)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Phase 1 Pharmacodynamic Study
MeSH Terms: interventions — salmon calcitonin; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1 Double Blind Oral rsCT Tablet (Experimental): Intervention: Oral rsCT tablet given once 4 hours after evening meal.
  Interventions: Drug: Oral rsCT tablet
- Part 1, Double-blind Oral Placebo Tablet (Placebo Comparator): Intervention: Oral placebo tablet matching the oral rsCT tablet, given once 4 hours after evening meal
  Interventions: Drug: Oral Placebo Tablet
- Part 2 Open label, Oral rsCT tablet (Experimental): Intervention: Oral rsCT tablet given once 2 hours after evening meal.
  Interventions: Drug: Oral rsCT tablet
- Part 2, Open Label Fortical Nasal Spray (Active Comparator): Intervention: Part 2 Open label. Fortical (rsCT) nasal spray given once 2 hours after evening meal
  Interventions: Drug: Fortical (rsCT) nasal spray

INTERVENTIONS:
Drug: Oral rsCT tablet — On Study Day 1, subjects will be given their assigned treatment, based on one of two randomly ordered treatment sequences, at 10 PM (22:00). On Visit 3, subjects will return for administration of the second treatment with a minimum of 7 days washout interval between study drug administrations. On Visit 4, subjects will return for administration of third treatment of rsCT, either oral rsCT tablets or Fortical (rsCT) nasal spray. Interventions are described in Intervention Name, Other Names and in Intervention Description.
  Other Names: rsCT
  Arms: Part 1 Double Blind Oral rsCT Tablet
Drug: Oral Placebo Tablet — Part 1, Double blind oral placebo tablet given once 4 hours after evening meal.
  Other Names: Placebo
  Arms: Part 1, Double-blind Oral Placebo Tablet
Drug: Oral rsCT tablet — Part 2, Open-label, oral rsCT tablet given once 2 hours after the evening meal.
  Arms: Part 2 Open label, Oral rsCT tablet
Drug: Fortical (rsCT) nasal spray — Intervention: Open label, Fortical nasal spray given once 2 hours after the evening meal.
  Other Names: Fortical nasal spray
  Arms: Part 2, Open Label Fortical Nasal Spray

SUMMARY:
This study is being conducted to assess the plasma CTx-1 concentrations when dosing is at night and to compare these results with those obtained with a placebo control and with commercially available nasal calcitonin.

DETAILED DESCRIPTION:
Timing of the dose of recombinant salmon calcitonin (rsCT) is important in effecting reduction of osteoclast activity. It is theorized that a dose administered before bedtime will be more effective than a dose administered in the morning. See protocol summary for information.

ELIGIBILITY:
Inclusion Criteria

* Postmenopausal female, in good health (at least five years since last menses).
* Age greater than or equal to 45 years old and less than or equal to 70 years old
* Weight ± 20% of the Metropolitan Life weight table.
* Plasma CTx-1 greater than or equal to 0.25 ng/ml.
* Total calcium, phosphorus, and magnesium within normal range.
* Willing and able to comply with all study requirements.
* Willing and able to sign written informed consent.
* Negative urine pregnancy test at screening.
* Negative Screen for Hepatitis B and C, HIV and drugs of abuse.

Exclusion Criteria:

* History of parathyroid, thyroid, pituitary or adrenal diseases.
* History of musculoskeletal disease.
* History of gastro-esophageal reflux disease (GERD) or other significant gastrointestinal disorders.
* History of cancer within 5 years of enrollment other than basal cell carcinoma.
* History of regular use of a Non-Steroidal Anti-inflammatory Drug (NSAID).
* History of surgery within 60 days of enrollment.
* History of hypersensitivity or allergies (other than seasonal allergies) within -years of enrollment including known sensitivity to the active ingredients or the excipients in the study medications.
* Use of concomitant medications other than acetaminophen within 7 days of enrollment or anticipated need to use such concomitant medications during the study.
* Use of bisphosphonates within 6 months, SERMS, estrogen or estrogen-like drugs 2 months, or calcitonin 1 month.
* Presence of any clinically significant illness.
* Unwilling or unable to comply with all study requirements.
* Unwilling or unable to sign written, informed consent.
* History of drug or alcohol abuse.
* Participation in any clinical study of an investigational drug within 60 days of enrollment.
* Plasma CTx-1 less than 0.25 ng/mL.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Legg, D.O., Principal Investigator — Bio-Kinetic Clinical Applications, Inc.
Locations (1):
- Bio-Kinetic Clinical Applications, Inc., Springfield, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Recombinant Salmon Calcitonin (rsCT): In Part 1, Period 1, 6 Subjects each were given rsCT tablets or 4 hours after the evening meal. In Part 1 Period 2, the same subjects were crossed over and given oral placebo 4 hours after the evening meal.
- Oral Placebo: In Part 1, Period 1, 6 Subjects each were given oral placebo tablets 4 hours after the evening meal. In Part 1 Period 2, the same subjects were crossed over and given oral rsCT tablets 4 hours after the evening meal.
- Oral rsCT Tablets (Part 2, Period 3): After completing Part 1, Periods 1 and 2, subjects were re-randomized to enter open label Part 2, Period 3, and received oral rsCT tablets given 2 hours after the evening meal.
- Fortical Nasal Spray (Part 2, Period 3): After completing Part 1, Periods 1 and 2, subjects were re-randomized to enter the open label Part 2, Period 3 and were given Fortical Nasal Spray 2 hours after the evening meal
Period: Part 1, Period 1
Arm/Group | Oral Recombinant Salmon Calcitonin (rsCT) | Oral Placebo | Oral rsCT Tablets (Part 2, Period 3) | Fortical Nasal Spray (Part 2, Period 3)
Started | 6 | 6 | 0 | 0
Completed | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Period 2
Arm/Group | Oral Recombinant Salmon Calcitonin (rsCT) | Oral Placebo | Oral rsCT Tablets (Part 2, Period 3) | Fortical Nasal Spray (Part 2, Period 3)
Started | 6 | 6 | 0 (No subjects were to be treated until after Periods 1 and 2.) | 0 (No subjects were to be treated until after Periods 1 and 2.)
Completed | 6 | 6 | 0 (No subjects treated.) | 0 (No subjects treated.)
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 3
Arm/Group | Oral Recombinant Salmon Calcitonin (rsCT) | Oral Placebo | Oral rsCT Tablets (Part 2, Period 3) | Fortical Nasal Spray (Part 2, Period 3)
Started | 0 (No subjects were treated in this period) | 0 (No subjects were treated in this period.) | 5 (Of the 6 eligible, 1 elected not to continue into Period 3.) | 4 (Of the 6 eligible, 2 elected not to continue into Period 3.)
Completed | 0 (No subjects were treated in this period) | 0 (No subjects were treated in this period.) | 5 (All who started this period completed) | 4 (All who started this period completed)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 12 women entered Part 1, the two-period crossover portion of the study; hence the same 12 received both oral treatments and should not be counted twice. Only 9 of those 12 went on to Part 2, the open label, non-crossover portion of the study.
Groups:
- Part 1 Oral rsCT Tablets: Subjects were given oral rsCT tablets 4 hours after the evening meal
- Part 1 Oral Placebo Tablets: Subjects were given oral placebo tablets 4 hours after the evening meal.
- Part 2 Open Label--Oral rsCT Tablets: After completing Part 1, Periods 1 and 2, subjects were eligible to participate in the open label Part 2 (Period 3) when oral rsCT tablets were given 2 hours after the evening meal.
- Part 2 Open Label Fortical Intranasal Spray: After completing Part 1, Periods 1 and 2, subjects were eligible to participate in the open label Part 2,(Period 3) when they received Fortical intra-nasal spray 2 hours after the evening meal
- Total: Total of all reporting groups
Arm/Group | Part 1 Oral rsCT Tablets | Part 1 Oral Placebo Tablets | Part 2 Open Label--Oral rsCT Tablets | Part 2 Open Label Fortical Intranasal Spray | Total
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (4.7) | 59.3 (4.7) |  |  | 59.3 (4.7)
Gender [Number; unit: participants]
  Female | 6 | 6 |  |  | 12
  Male | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 |  |  | 12
post-menopausal healthy females [Number; unit: participants] | 6 | 6 |  |  | 12
post-menopausal females [Number; unit: participants] | 6 | 6 |  |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic Effect of Oral Calcitonin
Description: C-terminal telopeptide of Collagen Type I (CTx-1) is an established plasma biomarker employed as an index of bone-resorption activity in response to interventions such as an anti-resorptive agent such as calcitonin. Here the calcitonin-salmon is rsCT, (recombinant) both oral and intranasal. These CTx-1 plasma concentrations were collected over 12 hours post-dosing where each subject served as her own control, as all received placebo in this crossover study, to account for the known diurnal variation of plasma CTx-1. For each time point, the ratio of the calcitonin response over the placebo response for that subject was derived from the plasma levels of CTx-1 and reported as a % of the placebo response (% Placebo or %P). These values were used to determine the primary pharmacodynamic parameter of Rmin, the minimum value seen following each active dose. The same %P values were used to derive the secondary pharmacodynamic parameters described in Secondary outc
Time Frame: 12 hr
Population: Not applicable. All participants who received treatment were included.
Measure: Mean (Standard Deviation); unit: percentage of time-matched placebo respo
Groups:
- Part 1 Oral rsCT Tablets: In this arm, Subjects were given oral rsCT tablets 4 hours after the evening meal.
- Part 1 Oral Placebo Tablets: In this arm, subjects were given oral placebo tablets 4 hours after the evening meal.
- Part 2 Oral rsCT Tablets: Subjects were given oral rsCT tablets four hours after the evening meal
- Part 2 Fortical Intra-nasal Spray: Subjects were given Fortical (rsCT) nasal spray four hours after the evening meal
Arm/Group | Part 1 Oral rsCT Tablets | Part 1 Oral Placebo Tablets | Part 2 Oral rsCT Tablets | Part 2 Fortical Intra-nasal Spray
Number analyzed (Participants) | 12 | 12 | 5 | 4
percentage of time-matched placebo respo | 37.5 (13.2) | 100 (NA) — As all values were converted to 100 percent, there was no variability | 41.2 (16.6) | 44.4 (21.8)

2. Secondary Outcome: Derived Pharmacodynamic Parameters Further Characterizing the Effects of Oral or Intranasal Calcitonin on Plasma CTx-1, Given at Night to Post-menopausal Women
Description: See Primary Outcome description. These CTx-1 plasma concentrations were collected over 12 hours, the values seen following active were compared with the time-matched individual values following placebo and used to derive the pharmacodynamic parameters. The primary was Rmin, seen above, and the Secondary ones were the time to that Rmin (Tmin) and the total time from the beginning of the inhibition to the end of the effect or the end of the study period (Tinhibition).
Time Frame: 12 hours
Population: Data from Part 1 (crossover Periods 1 and 2) were pooled to give CTx-1 mean data for the oral rsCT tablet group (n = 12) and for the oral placebo group n = 12). Part 2, open-label, non-crossover, compared the CTx-1 results after oral rsCT (n = 5) with those after Fortical(n = 4. The % inhibition is reported first.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Part 2 Oral rsCT Tablets: After completing Part 1, subjects were eligible to enter the open-label Part 2. One dropped out and 5 entered and received oral rsCT tablets given 2 hours after the evening meal.
- Part 2 Fortical Intra-nasal Spray: After completing Part 1, subjects were eligible to enter the open-label Part 2. Two dropped out and 4 received Fortical nasal spray 2 hours after the evening meal.
Arm/Group | Part 1 Oral rsCT Tablets | Part 1 Oral Placebo Tablets | Part 2 Oral rsCT Tablets | Part 2 Fortical Intra-nasal Spray
Number analyzed (Participants) | 12 | 12 | 4 | 5
Hours
  Tmin=time in hours to Rmin | 7.5 (5.0) | 0 (0) | 4.5 (5.0) | 4.0 (3.5)
  TInhibition=total time of effect in hours | 10.9 (2.0) | 0 (0) | 9.9 (2.6) | 10.7 (3.0)

3. Secondary Outcome: AUCInhibition=Hours*%P
Description: The AUCinhibition, (Area Under the Inhibition Curve) in hours*%inhibition vs placebo under the baseline line over the curve.
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: hours*%P
Arm/Group | Part 1 Oral rsCT Tablets | Part 1 Oral Placebo Tablets | Part 2 Oral rsCT Tablets | Part 2 Fortical Intra-nasal Spray
Number analyzed (Participants) | 12 | 12 | 4 | 5
hours*%P | 474.7 (267.7) | 0 (0) | 345.8 (279.0) | 504.7 (477.4)

ADVERSE EVENTS:
Time Frame: Any time within the treatment period up to 30 days after treatment
Arm/Group | Part 1 Oral rsCT Tablets | Part 1 Oral Placebo Tablets | Part 2 Open Label--Oral rsCT Tablets | Part 2 Open Label Fortical Intranasal Spray
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/12 | 3/12 | 0/5 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Oral rsCT Tablets (N=12) | Part 1 Oral Placebo Tablets (N=12) | Part 2 Open Label--Oral rsCT Tablets (N=5) | Part 2 Open Label Fortical Intranasal Spray (N=4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
eyelid edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except as provided herein or as required by applicable law, you agree that you shall keep such Unigene Information confidential and that you shall not, without our prior written consent, transmit, publish, or otherwise disclose to any person or entity either (i) the Unigene Information, (ii) the fact of our disclosure of the Unigene Information to you, or (iii) the existence or terms of any negotiations or discussions between us regarding your potential engagement.